CLINICAL TRIAL: NCT07118475
Title: Exploratory Clinical Study of Adult Pancreatic Progenitor-derived Islet Autologous Transplantation in the Treatment of Diabetes
Brief Title: Autologous Islet Transplantation for Diabetes
Acronym: APPITD
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-257
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2)
Keywords: diabetes; islet transplantation; adult pancreatic progenitor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous islet transplantation (Experimental)
  Interventions: Biological: Autologous islet transplantation

INTERVENTIONS:
Biological: Autologous islet transplantation — 1. EUS-FNB or surgical procurement of pancreatic tissue
  2. In vitro culture of adult pancreatic progenitor
  3. In vitroinduction of islets
  4. islet transplantation beneath the anterior rectus sheath
  5. Post-transplant follow-up

SUMMARY:
This study aims to conduct an exploratory clinical trial recruiting insulin-dependent diabetic patients who meet the criteria for islet transplantation. Pancreatic tissue will be obtained via endoscopic ultrasound-guided fine-needle aspiration biopsy, and adult pancreatic progenitor cells (APP) will be expanded in vitro and differentiated into islet-like cells. After quality assessment, these cells will be transplanted via injection beneath the anterior rectus sheath.

Following autologous transplantation of APP-derived islets, the transplanted islets are expected to survive at the implantation site, stably secrete insulin, and thereby reduce or potentially eliminate the need for exogenous insulin. Glycated hemoglobin (HbA1c) levels are anticipated to decrease, with a significant reduction in the risk of severe hypoglycemic episodes, and no transplant-related adverse events are expected.

As this is an exploratory clinical study, participants may not benefit from APP islet transplantation and may face risks or adverse events associated with the procedure. However, the findings of this research may advance more scientific and effective treatment strategies for diabetes. The successful completion of this study could provide a feasible and scalable approach to functionally curing diabetes, effectively reducing disability and mortality rates among diabetic patients, improving their quality of life, and generating substantial health, economic, and social benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients with islet transplantation indications
2. Dependent on exogenous insulin therapy
3. C-peptide <0.3 ng/ml or blood glucose control remains unsatisfactory despite intensive insulin therapy.

Exclusion Criteria:

1. Unable to tolerate transplant related procedures for various reason
2. Persons with a history of infectious diseases such as hepatitis B, hepatitis C, HIV and tuberculosis, or persons with active bacterial, fungal or viral infection
3. Heart, liver and kidney dysfunction or significant decrease in blood cells
4. Previous cancer history
5. Researcher-deemed ineligible for this clinical trial due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Within one year after transplant
  Adverse events will be coded according to the MedDRA dictionary, and AE will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 of the National Cancer Institute.
Hypoglycemia incidence rate | Within one year after transplant
  Hypoglycemia can be divided into three levels based on blood sugar levels, physical changes, and state of consciousness.

SECONDARY OUTCOMES:
Changes in glycosylated hemoglobin (HbA1c) from baseline at 3 months, 6 months, 9 months, and 1 year after transplantation | Within one year after transplant
  Changes in glycosylated hemoglobin (HbA1c) from baseline at 3 months, 6 months, 9 months, and 1 year after transplantation
Changes in time in range (TIR) at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline | Within one year after transplant
  The changes in time in range (TIR) at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline.
Changes in fasting plasma glucose at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline | Within one year after transplant
  The changes in fasting plasma glucose at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline
Changes in insulin at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline | Within one year after transplant
  The changes in insulin level at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline
Changes in C-peptide at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline | Within one year after transplant
  The changes in C-peptide level at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline
Changes in exogenous insulin dosage at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline | Within one year after transplant
  Changes in exogenous insulin dosage at 3 months, 6 months, 9 months, and 1 year post-transplantation compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Lin, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form and clinical study report will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From study publication to 5 years post-study
Access Criteria: For academic inquiries or research collaboration, interested investigators may contact the Principal Investigator, Professor Shengli Lin, via email.
URL: https://clinicaltrials.gov